CLINICAL TRIAL: NCT00545896
Title: Safety and Efficacy Study for the Use of Extracorporeal Shockwaves in the Treatment of Chronic Soft Tissue Wounds
Brief Title: Extracorporeal Shockwave Treatment for Chronic Soft Tissue Wounds
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AUVA (Other)
Responsible Party: Wolfgang SCHADEN, MD, UKH Meidling - AUVA
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESWT 001 - 2003
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2009-08

CONDITIONS: Chronic Nonhealing Wounds
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Extracorporeal shockwave therapy — Extracorporeal application of shockwaves on the surface of chronic wounds.

SUMMARY:
Chronic soft tissue wounds represent a difficult problem for patients and doctors as well. Chronic wounds can be caused by internal and dermatological diseases like venous ulcers as a consequence of venous insufficiency, arterial ulcers as a consequence of peripheral occlusive vascular disease, the diabetic foot stemming from diabetes and other pathologies. A different reason for chronic wounds could be prior traumatic injuries (war wounds, traffic accidents)not showing a tendency to heal after surgical repair.

The primary goal in the treatment of chronic soft tissue wounds is to obtain wound closure. Usually necrotic tissue is debrided, i.e. surgically removed, to assess the full extent of the damage, to detect underlying abscesses or other pathologies causing the non-healing of the wound. Wet - to - wet dressings are primarily applied to induce a healing process. As second line attempts to obtain closure special dressings like semipermeable films, gels, hydrocolloids and calcium alginates are applied. These expensive dressings are associated with extended time periods of conservative treatment until closure can be observed.

A third line after failure of nonoperative treatment is the application of skin graft. This involves the operative and anesthesiological risk for an already health wise compromised patient with little to no physiological reserve. One should not forget that the majority of patients presenting at outpatient clinics with chronic soft tissue wounds are the elderly with/without disabling comorbidities.

The use of extracorporeal shockwaves (ESW) for clinical applications was introduced in central Europe more than two decades ago. Extracorporeal shockwave therapy (ESWT)is used in the fields of urology, orthopedic surgery, trauma surgery. ESW are associated with the induction of neovascularisation and with mechanical stimuli causing proliferation of a large number of cells including osteoblasts (Martini L., J Trauma 2006). The exact effects of ESW on human cells are currently studied in several centers worldwide. The application of ESWT in the above mentioned fields of medicine proved safe, reliable and almost complication-free.

Our center's experience with ESWT in trauma surgery (Schaden W., Clin. Orthop 2001)and the observation that not only the traumatic condition (fracture non-union, etc.), but also the surrounding tissue showed favorable tissue healing after ESWT, leads to our hypothesis that ESWT might be beneficial for the much larger number of chronic soft tissue wounds. The investigators anticipate to induce complete wound healing in a number of defined clinical/pathological conditions by ESWT. At the same time efficacy and safety of ESWT will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a chronic soft tissue wound persisting for longer than one month.
* Cause of chronic wound irrelevant except circumferential second degree burn wounds of upper/lower extremity.
* Capable of wound care at home or home nursing available.
* Patients older than 18 years.
* The patient is willing, able to read, understand and willing to give informed consent to the study procedure.
* Female patients will not be pregnant.
* The patient will agree to an outpatient clinic treatment.
* The patient agrees to comply with the protocol requirements, including the self care of wounds and all follow up visit requirements

Exclusion Criteria:

* Pregnancy
* Active or previous (within 8 weeks to the study screening visit) chemotherapy
* Deep vein thrombosis within 6 months to the study screening visit
* Lower extremity revascularization procedure (e. g. PTA, graft or other) within 8 weeks to the study screening visit
* Current history of substance abuse
* Physical or mental disability ( if not cared for, i. e. home nursing etc)or geographical concerns (residence not within reasonable travel distance to study center)that would hamper compliance with required study visits
* Current participation in another clinical investigation of a medical device or a drug, or recent participation in such a study within 8 weeks to the study screening visit
* The investigator believes that the subject will be unwilling or unable to comply with the study protocol requirements, including the ESWT procedure, standard of care self-care requirements and all study related follow-up visit requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2003-09; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 30 days after last ESWT session

SECONDARY OUTCOMES:
Rate of complete wound closure and number of ESWT sessions needed. Rate of nonhealing wounds and number of ESWT sessions until drop out/ reasons for drop out. | 30 days after last ESWT session or drop out date.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus S. WOLFF, MD, Principal Investigator — Heeresspital - Wien - Austrian Armed Forces Hospital - Vienna
Locations (1):
- Unfallkrankenhaus Meidling - Trauma Center Meidling, Vienna, Austria

REFERENCES:
- [Result] Wolff KS, Wibmer A, Pusch M, Prusa AM, Pretterklieber M, Teufelsbauer H, Schaden W. The influence of comorbidities and etiologies on the success of extracorporeal shock wave therapy for chronic soft tissue wounds: midterm results. Ultrasound Med Biol. 2011 Jul;37(7):1111-9. doi: 10.1016/j.ultrasmedbio.2011.04.007. Epub 2011 Jun 2. PMID 21640475